CLINICAL TRIAL: NCT02282813
Title: A Long-term Safety and Efficacy Study of CTAP101 Capsules in Subjects With Stages 3 or 4 Chronic Kidney Disease, Secondary Hyperparathyroidism and Vitamin D Insufficiency (Extension of Study CTAP101-CL-3001 or CTAP101-CL-3002)
Brief Title: Extension Study of CTAP101-CL-3001 or CTAP101-CL-3002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTAP101-CL-3003
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Kidney Disease; Hyperparathyroidism, Secondary; Vitamin D Deficiency
Keywords: Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism, Secondary; Vitamin D; Hyperparathyroidism; Kidney Diseases; Kidney Failure; Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Vitamin D Deficiency; Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism; Kidney Diseases | interventions — Calcifediol; Calcitriol; 1 alpha-hydroxyergocalciferol; paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CTAP101 Capsules alone (Experimental): CTAP101 Capsules 30 or 60 mcg daily for up to 26 weeks
  Interventions: Drug: CTAP101 Capsules
- CTAP101 Capsules +calcitriol (Experimental): CTAP101 Capsules 60 mcg +calcitriol daily for 14 weeks
  Interventions: Drug: CTAP101 Capsules; Drug: Calcitriol
- CTAP101 Capsules +doxercalciferol (Experimental): CTAP101 Capsules 60 mcg +doxercalciferol daily for 14 weeks
  Interventions: Drug: CTAP101 Capsules; Drug: Doxercalciferol
- CTAP101 Capsules +paricalcitol (Experimental): CTAP101 Capsules 60 mcg +paricalcitol daily for 14 weeks
  Interventions: Drug: CTAP101 Capsules; Drug: Paricalcitol

INTERVENTIONS:
Drug: CTAP101 Capsules — At week 12, eligible subjects will continue to take 1-2 capsules (30 mcg each capsule) CTAP101 daily
  Other Names: Calcifediol
Drug: Calcitriol — At week 12, eligible subjects will be randomized to also take calcitriol 0.25 mcg dose one capsule daily
  Other Names: calcifediol
  Arms: CTAP101 Capsules +calcitriol
Drug: Doxercalciferol — At week 12, eligible subjects will be randomized to also take doxercalciferol 0.5 mcg one capsule daily
  Other Names: calcifediol
  Arms: CTAP101 Capsules +doxercalciferol
Drug: Paricalcitol — At week 12, eligible subjects will be randomized to also take paricalcitol 1 mcg one capsule daily
  Other Names: calcifediol
  Arms: CTAP101 Capsules +paricalcitol

SUMMARY:
This extension study of subjects previously enrolled in studies CTAP101-CL-3001 or CTAP101-CL-3002 allows long term evaluation of the safety and efficacy of CTAP101 Capsules in reducing elevated intact parathyroid hormone (iPTH) and correcting vitamin D insufficiency in stage 3 or 4 chronic kidney disease patients.

DETAILED DESCRIPTION:
Only subjects previously enrolled in studies CTAP101-CL-3001 or CTAP101-CL-3002 are eligible to participate in this extension study. This is a phase 3, open-label study of CTAP101 Capsules, with and without add-on vitamin D hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Completed either of the phase 3 double-blind, placebo-controlled studies, CTAP101-CL-3001 or CTAP101-CL-3002
* Taking no more than 1000 mg/day of elemental Ca and willing/able to remain on this dose for the duration of the study
* Taking no more than 1600 IU/dose vitamin D (ergocalciferol or cholecalciferol) therapy and willing/able to remain on a stable dose of vitamin D during the study
* Willing and able to comply with study instructions and to commit to all clinic visits for the duration of the study
* Female subjects of childbearing potential must be neither pregnant nor lactating and must have a negative urine pregnancy test
* All female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use effective contraception (eg, implants, injectables, combined oral contraceptives, intrauterine device, sexual abstinence, vasectomy or vasectomized partner) for the duration of the study
* Have the ability to read and understand subject Informed Consent Form (ICF). Subjects or their legal representatives must sign the ICF.

Exclusion Criteria:

* Use of pharmacological dose of ergocalciferol and cholecalciferol (monthly equivalent of 50,000 IU or 1250 µg, eg, Drisdol®) or bisphosphonate therapy
* Use of other bone metabolism therapy (with the exception of stable doses of bisphosphonates and denosumab [Xgeva® and Prolia®]) that may interfere with study endpoints
* Concomitant serious illness or medical condition, such as malignancy, human immunodeficiency virus, significant gastrointestinal or hepatic disease or cardiovascular event or hepatitis that in the opinion of the investigator may worsen and/or interfere with participation in the study
* Neurological/psychiatric disorder, including psychotic disorder or dementia, or any condition reason which, in the opinion of the investigator makes adherence to a treatment or follow-up schedule unlikely
* Known or suspected hypersensitivity to any of the constituents of either investigational product (CTAP101) or adjunctive vitamin D hormone therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Melnick, MD, Study Director — OPKO Renal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects could enroll in extension study after completing trials CTAP101-CL-3001 or CTAP101-CL-3002. Subjects from 68 sites participated with at least 1 subject enrolled in the extension per site. Three sites participated in both blinded trials.
Pre-assignment Details: Treatment groups were categorized as treated for 26 weeks; subjects previously on placebo in predecessor trials) or 12 months (52 weeks; subjects previously on active treatment in predecessor trials). Following 12 weeks, a subset of eligible subjects (n=up to 90) could be randomized to take adjunctive therapy in addition to CTAP101 capsules.
Groups:
- CTAP101 Capsules (Not Randomized; 6 Mos Treatment): CTAP101 Capsules 30 or 60 mcg daily for up to 12 weeks, followed by additional weeks 13-26.
  CTAP101 Capsules: At end of week 12, eligible subjects will continue to take 1 or 2 capsules (30 mcg each capsule) CTAP101 daily.
- CTAP101 Capsules (Not Randomized; 12 Mos Treatment): CTAP101 Capsules 30 or 60 mcg daily for up to 12 weeks followed by additional weeks 13-26.
  CTAP101 Capsules: At end of week 12, eligible subjects will continue to take 1 or 2 capsules (30 mcg each capsule) CTAP101 daily
- CTAP101 Caps 2 x 30 mcg Daily for 12 wk+Adjunctive: CTAP101 Capsules 2 x 30 mcg daily for up to 12 weeks. At week 12, a subset of eligible subjects (N=85) were randomized to take adjunctive therapy (calcitriol 0.25 mcg or doxercalciferol 0.5 mcg or paricalcitol 1 mcg) daily in addition to the CTAP101 capsules.
Period: Overall Study
Arm/Group | CTAP101 Capsules (Not Randomized; 6 Mos Treatment) | CTAP101 Capsules (Not Randomized; 12 Mos Treatment) | CTAP101 Caps 2 x 30 mcg Daily for 12 wk+Adjunctive
Started | 103 (ITT Population) | 153 (ITT Population - not randomized or randomized to CTAP101 monotherapy) | 42 (Randomization to take adjunctive treatment in addition to CTAP101 capsules began after week 12.)
Completed | 91 | 130 | 39
Not Completed | 12 | 23 | 3
Not completed — Withdrawal by Subject | 4 | 5 | 0
Not completed — Adverse Event | 3 | 10 | 1
Not completed — Subject non-compliance | 1 | 4 | 0
Not completed — Physician Decision | 0 | 3 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Serum Ca >/=11.0mg/dL | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Administrative reasons | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population: includes subjects receiving CTAP101 capsules only in the extension trial (up to 6 months total active therapy, subjects receiving up to 12 months receiving CTAP101 capsules (6 months in the previous trials and up to 6 months in the extension) with or without being randomized to CTAP101 capsules plus adjunctive therapy.
Groups:
- CTAP101 Capsules (Monotherapy; 12 Mos Treatment): CTAP101 Capsules 30 or 60 mcg daily for up to 12 weeks followed by additional weeks 13-26.
  CTAP101 Capsules: At end of week 12, eligible subjects will continue to take 1 or 2 capsules (30 mcg each capsule) CTAP101 daily
- Total: Total of all reporting groups
Arm/Group | CTAP101 Capsules (Not Randomized; 6 Mos Treatment) | CTAP101 Capsules (Monotherapy; 12 Mos Treatment) | CTAP101 Caps 2 x 30 mcg Daily for 12 wk+Adjunctive | Total
Number analyzed (Participants) | 103 | 153 | 42 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.78) | 66.9 (9.83) | 65.0 (12.34) | 65.9 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 85 | 14 | 154
  Male | 48 | 68 | 28 | 144
Region of Enrollment [Number; unit: participants]
  United States | 103 | 153 | 42 | 298

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in the Intent to Treat Population With a Mean Reduction in Plasma Intact Parathyroid Hormone (iPTH) of >/= 30% From Baseline Values at End of Treatment (EOT)
Description: Number of subjects in the intent to treat population with a mean reduction in plasma intact parathyroid hormone (iPTH) of >/= 30% from pretreatment baseline values at end of treatment (EOT), classified as responders
Time Frame: up to 6 months
Population: Intent to treat
Measure: Number; unit: participants
Groups:
- CTAP101 Capsules (Not Randomized; 6 Mos Treatment): CTAP101 Capsules 30 or 60 mcg daily for up to 12 weeks, followed by additional weeks 13-26.
  CTAP101 Capsules: At end of week 12, eligible subjects continued to take 1 or 2 capsules (30 mcg each capsule) CTAP101 daily.
- CTAP101 Capsules (Not Randomized; 12 Mos Treatment): CTAP101 Capsules 30 or 60 mcg daily for up to 12 weeks followed by additional weeks 13-26.
  CTAP101 Capsules: At end of week 12, eligible subjects continued to take 1 or 2 capsules (30 mcg each capsule) CTAP101 daily
Arm/Group | CTAP101 Capsules (Not Randomized; 6 Mos Treatment) | CTAP101 Capsules (Not Randomized; 12 Mos Treatment) | CTAP101 Caps 2 x 30 mcg Daily for 12 wk+Adjunctive
Number analyzed (Participants) | 103 | 153 | 42
participants | 34 | 66 | 30
Statistical Analysis 1: Comparison: CTAP101 Capsules (Not Randomized; 6 Mos Treatment) vs CTAP101 Capsules (Not Randomized; 12 Mos Treatment); Test type: Superiority or Other; p = 0.1041, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Participants in the Per Protocol Population With Mean Reduction in Plasma Intact Parathyroid Hormone (iPTH) of >/= 30% From Baseline Values at End of Treatment (EOT)
Description: Number of subjects in the per protocol population with a mean reduction in plasma intact parathyroid hormone (iPTH) of >/= 30% from pretreatment baseline values at end of treatment (EOT), classified as responders
Time Frame: up to 6 months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | CTAP101 Capsules (Not Randomized; 6 Mos Treatment) | CTAP101 Capsules (Not Randomized; 12 Mos Treatment) | CTAP101 Caps 2 x 30 mcg Daily for 12 wk+Adjunctive
Number analyzed (Participants) | 91 | 126 | 40
participants | 34 | 64 | 29
Statistical Analysis 1: Comparison: CTAP101 Capsules (Not Randomized; 6 Mos Treatment) vs CTAP101 Capsules (Not Randomized; 12 Mos Treatment); Test type: Superiority or Other; p = .0503, Cochran-Mantel-Haenszel

3. Secondary Outcome: Number of Participants in the Intent to Treat Population With Normal Serum 25-hydroxyvitamin D at End of Treatment (EOT)
Description: Number of Participants in the Intent to Treat Population with serum 25-hydroxyvitamin D >/= 30 ng/mL at End of Treatment (EOT)
Time Frame: up to 6 months
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | CTAP101 Capsules (Not Randomized; 6 Mos Treatment) | CTAP101 Capsules (Not Randomized; 12 Mos Treatment) | CTAP101 Caps 2 x 30 mcg Daily for 12 wk+Adjunctive
Number analyzed (Participants) | 103 | 153 | 42
participants | 87 | 124 | 38
Statistical Analysis 1: Comparison: CTAP101 Capsules (Not Randomized; 6 Mos Treatment) vs CTAP101 Capsules (Not Randomized; 12 Mos Treatment); Test type: Superiority or Other; p = 0.4817, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Participants in the Per Protocol Population With NormalSerum 25-hydroxyvitamin D at End of Treatment (EOT)
Description: Number of Participants in the per protocol population with serum 25-hydroxyvitamin D >/= 30 ng/mL at End of Treatment (EOT)
Time Frame: up to 6 months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | CTAP101 Capsules (Not Randomized; 6 Mos Treatment) | CTAP101 Capsules (Not Randomized; 12 Mos Treatment) | CTAP101 Caps 2 x 30 mcg Daily for 12 wk+Adjunctive
Number analyzed (Participants) | 91 | 126 | 40
participants | 86 | 120 | 37
Statistical Analysis 1: Comparison: CTAP101 Capsules (Not Randomized; 6 Mos Treatment) vs CTAP101 Capsules (Not Randomized; 12 Mos Treatment); Test type: Superiority or Other; p = 0.8086, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 6 months from initiation of treatment through end of treatment
Arm/Group | CTAP101 Capsules (Not Randomized; 6 Mos Treatment) | CTAP101 Capsules (Not Randomized; 12 Mos Treatment) | CTAP101 Caps 2 x 30 mcg Daily for 12 wk+Adjunctive
Serious Adverse Events (participants affected / at risk) | 18/103 | 33/153 | 9/42
Other Adverse Events (participants affected / at risk) | 36/103 | 54/153 | 22/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTAP101 Capsules (Not Randomized; 6 Mos Treatment) (N=103) | CTAP101 Capsules (Not Randomized; 12 Mos Treatment) (N=153) | CTAP101 Caps 2 x 30 mcg Daily for 12 wk+Adjunctive (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eschericia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eschericia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood creatinine phosphokinase MB increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal ganglia inferction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglcaemic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTAP101 Capsules (Not Randomized; 6 Mos Treatment) (N=103) | CTAP101 Capsules (Not Randomized; 12 Mos Treatment) (N=153) | CTAP101 Caps 2 x 30 mcg Daily for 12 wk+Adjunctive (N=42)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 9 (9) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (7) | 6 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 5 (5) | 2 (2)
Oedema peripheral (General disorders) | 6 (6) | 5 (5) | 0 (0)
Fatigue (General disorders) | 7 (7) | 3 (3) | 1 (1)
Urinary tract obstruction (Infections and infestations) | 2 (2) | 10 (10) | 1 (1)
Gout (Metabolism and nutrition disorders) | 7 (7) | 2 (2) | 1 (1)
Oedema (General disorders) | 2 (2) | 2 (2) | 3 (3)
Blood creatinine increased (Investigations) | 3 (3) | 6 (6) | 3 (3)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 4 (4) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less